CLINICAL TRIAL: NCT04647474
Title: A Prospective and Longitudinal Cohort Study Assessing Mental wellbeIng and Quality of Life in Prostate Cancer - the MIND-P Study
Brief Title: Mental Wellbeing and Quality of Life in Prostate Cancer
Acronym: MIND-P
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: King's College Hospital NHS Trust (Other); Guy's and St Thomas' NHS Foundation Trust (Other); Imperial College Healthcare NHS Trust (Other); Medway NHS Foundation Trust (Other); Lewisham and Greenwich NHS Trust (Other Government); Surrey and Sussex Healthcare NHS Trust (Other); Bedfordshire Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 284473
Record Dates: First submitted 2020-11-23; First posted 2020-12-01 (Actual); Last update posted 2023-05-26 (Actual); Status verified 2023-05

CONDITIONS: Prostate Cancer
Keywords: Prostate Cancer; Depression; Anxiety; Mental Wellbeing; Functional Outcomes; Social Wellbeing
MeSH Terms: conditions — Prostatic Neoplasms; Depression; Anxiety Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Radical Prostatectomy: Participants undergoing any curative surgical treatment option for prostate cancer irregardless of approach (open, laparoscopic or robotic)
- Active Surveillance: Participants undergoing active surveillance as the management option for prostate cancer as defined by regular surveillance attendance at the primary treating site.
- Hormone Monotherapy: Participants undergoing medical hormone therapy (Antiandrogens and Gonadotropin-releasing hormone (GnRH) agonists or antagonists) or surgical castration (e.g. orchidectomy) options as the primary treatment for prostate cancer.
- Radical Radiotherapy: Participants undergoing primary radiotherapy treatment for prostate cancer irregardless of delivery methods (e.g. External beam radiation therapy or brachytherapy).

SUMMARY:
The complex relationship that exists between physical and mental health in prostate cancer is increasingly being understood. Psychiatric symptoms are common in this group and have important consequences for the quality of life and cancer outcomes for patients with prostate cancer. However, less is understood about the severity of disease and which patient factors and treatment options are risk factors for developing problems. Additionally, the impact these conditions have on problems such as urinary incontinence or sexual function is less well understood. The investigators anticipate that different patient characteristics and treatment options increase an individuals risk of developing problems after a prostate cancer diagnosis. Therefore, this study aims to further investigate these specific factors to improve follow up care in patients with prostate cancer.

This observational study will follow up newly diagnosed prostate cancer patients for a period of 12 months to evaluate these outcomes. Participants will be identified across seven hospitals in London and South England. After being recruited participants will be invited to undergo repeated online or postal questionnaires at baseline, 3, 6, 9 and 12 months. These will assess depressive and anxiety symptom load, body image issues, fear of recurrence, masculinity perception and functional symptoms (including urinary, bowel and sexual symptoms) load.

Analysis of these findings will allow for identification of 1) Which subgroups of patients appear to have worse mental wellbeing and quality of life outcomes, and 2) How mental health issues impact functional outcomes. This will provide important information for guiding future research within the subject area and further inform clinicians about these issues.

DETAILED DESCRIPTION:
Prostate cancer represents a large proportion of global cancer incidence, accounting for 13.5% of all male cancers. However, with high survival rates, which are still improving, there is growing acceptance that living longer does not always equate to living well. The mental health aspect of the disease is unfortunately sometimes neglected with research focusing on the physical symptoms after disease much more prominent and frequently conducted. Previous research has already demonstrated that mental health issues are common in patient with prostate cancer, however, less is known about which patients are at greater risk of developing problems after being diagnosed with prostate cancer. Additionally, the association between mental health conditions and what are called 'functional outcomes' (i.e. bladder, bowel and sexual function) after treatment are less well understood. A greater knowledge of these factors can help clinicians to make better assessments of patients and also will help the future development of additional tools which are able to help with diagnosis in future.

With these factors in mind the primary aims of the research study is :

1. To evaluate the association between prostate cancer patients undergoing different treatments and overall mental wellbeing in the initial cancer follow-up stage.

The secondary aims of the study are to:

1. Identify high risk time-frames post diagnosis for worsening of mental wellbeing
2. Assess the impact of depressive and anxiety symptoms on functional, clinical and other mental wellbeing outcomes.
3. Explore patient and cancer related factors conferring a risk for the development of significant mental wellbeing problems.

The investigators hypothesis is that prostate cancer patients experience a high psychological symptom load in the initial follow up period after diagnosis. Additionally, based on previous prostate cancer and mental health research the investigators hypothesise that certain subgroups (e.g. certain treatment or patient groups) are at increased risk of developing significant psychological symptoms.

To explore these aims and hypothesis the investigators will conduct a questionnaire based, longitudinal and observational cohort study of participants recently diagnosed with prostate cancer. There is no interventional element to the study. The investigators will identify newly diagnosed patients, who have not yet received treatment from multiple hospital sites in London and the South East of England. This will include patients allocated to surgery, radiotherapy, surveillance or hormone therapy depending on prostate cancer characteristics. Participants will be identified by the clinical team during the hospital outpatient appointment, with contact details taken at this stage. The investigators are aiming to recruit 300 participants for this study based on power calculations (80% power with 0.05 significance) for the primary outcomes taking into account a maximum drop out rate of 25%.

Following identification, screening and consenting for inclusion into the study participants will begin data collection through serial questionnaires. Participants will have the option of either undergoing postal or electronic follow up, depending on preference. Questionnaires will include numerous validated measures to evaluate mental and social wellbeing as well as functional symptoms of disease/treatment including bladder, bowel and sexual function as per the outcome measures described.

Collection of data will occur at set intervals for the duration of the study and will include the same questionnaire being filled at the beginning of the study, 3, 6, 9 and 12 months. Additionally, at the outset of the study some further information will be asked from the participant including demographics and previous medical or psychiatric history. The research team will in addition collect data from the medical files at the beginning of the study about the cancer characteristics and then again at the end of the study at 12 months. At 12 months participants will complete the study and data analysis along the primary and secondary outcome measures will be conducted once all participants have completed this.

ELIGIBILITY:
Inclusion Criteria:

* New diagnosis of histologically proven or clinically likely prostate cancer

  * No limits on grade, histology type or risk stratification classification
* Post Multi Disciplinary Team discussion with allocation of a suggested treatment or follow up strategy
* Undergoing one of the following four treatment/management options:

  * Radical Prostatectomy
  * Radiotherapy (External beam radiation therapy or brachytherapy)
  * Active Surveillance
  * Androgen Deprivation Therapy (Medical or Surgical castration)
* Follow up undertaken by urology, oncology or mixed uro-oncology teams

Exclusion Criteria:

* Patient is pre-Multi Disciplinary Team discussion
* Patient has already undergone the allocate intervention

  * Post-surgery
  * Post first radiotherapy dose
  * Attended second active surveillance follow up
  * Received >1 dose (initial dose) of Gonadotropin-releasing hormone agonist/antagonist
* Patients receiving the following therapies:

  * Palliative patients on symptom control only
  * Patients allocated to watchful waiting
  * Any type of Focal therapy e.g. high intensity focused ultrasound (HIFU)
  * Patients receiving adjuvant combination therapy e.g. Androgen deprivation therapy or chemotherapy pre radiotherapy or surgery
  * Metastatic patients undergoing chemotherapy alone
* Patients presenting with recurrence or progression of prostate cancer
* Concurrent management for another cancer diagnosis
* Recent admission to an inpatient psychiatric facility within the previous 12 months prior to diagnosis of prostate cancer
* Patients lacking capacity to consent or undertake in the research
* Those unable to complete the required surveys, such as those not able to understand English or those with severe learning disability

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population of study are patients with a recently newly confirmed diagnosis, or clinically likely diagnosis of prostate cancer in a secondary care setting. Four separate sub-cohorts based on treatment or management allocated will be recruited with identical inclusion and exclusion criteria, with the exception of treatment specific characteristics. The four cohorts to be recruited will be newly diagnosed men with prostate are those described in the eligibility criteria.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-03-29 (Actual); Study Completion 2023-03-29 (Actual)

PRIMARY OUTCOMES:
Mean difference of mental wellbeing measures between four management groups | Baseline, 3, 6, 9 and 12 months post diagnosis
  Mental wellbeing validated tools scores including Patient Health Questionnaire-9 (PHQ-9), Generalised Anxiety Disorder-7 (GAD-7), Body Image Scale, Fear of Recurrence Scale and Masculine Self-Esteem Prostate Cancer-Related Quality of Life (PC-QOL) Subset Scale

SECONDARY OUTCOMES:
Cumulative incidence of significant mental wellbeing outcomes | 12 Months
  Binary outcome of the development of significant individual mental wellbeing outcomes (depression, anxiety, body image issues, masculinity and fear of cancer recurrence)
Exploration of prognostic factors of mental wellbeing outcomes. | Within 12 months of diagnosis
  Pre-selected patient, oncological and treatment factors evaluated against each individual mental wellbeing outcome for exploration of potentially prognostic factors for significant symptom development.
Relationship between each individual mental wellbeing symptom and functional/social wellbeing. | At 12 months post diagnosis.
  Functional outcomes will include sexual, urinary and bowel symptoms from EPIC-26. Social wellbeing will include FACT-G subscale scores with general health defined using the SF-12 physical component score.
Evaluation of effect of time on symptoms | Within 12 months of diagnosis
  Evaluate the trajectory of mental wellbeing symptoms over a 12-month period and effect of time on symptom scores.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran Ahmed, MBBS, FRCS, Principal Investigator — King's College London
Locations (7):
- United Kingdom (7):
  - Bedfordshire Hospitals NHS Foundation Trust, Bedford, Bedfordshire
  - Guy's and St Thomas' NHS Foundation Trust, London, Greater London
  - Lewisham and Greenwich NHS Trust, London, Greater London
  - King's College Hospital NHS Foundation Trust, London, Greater London
  - Imperial College Healthcare NHS Trust, London, Greater London
  - Medway NHS Foundation Trust, Gillingham, Kent
  - Surrey and Sussex Healthcare NHS Trust, Redhill, Surrey

IPD SHARING:
Plan to Share IPD: Yes
Anonymised individual participant data pertaining to any analysis conducted by this research will be made available publicly without restriction after the conductance of the study through the King's Research Data Repository.
Supporting Information: SAP, Analytic Code
Time Frame: All raw data will be made available by the time of publication of the research study in a peer reviewed journal. This will be archived for a duration of 20 years.
Access Criteria: Openly available through the King's Research Data Repository.

REFERENCES:
- [Derived] Brunckhorst O, Liszka J, James C, Fanshawe JB, Hammadeh M, Thomas R, Khan S, Sheriff M, Muir G, Ahmed HU, Van Hemelrijck M, Stewart R, Dasgupta P, Ahmed K. Mental well-being in prostate cancer: A multi-institutional prospective cohort study. BJUI Compass. 2025 Jun 17;6(6):e70040. doi: 10.1002/bco2.70040. eCollection 2025 Jun. PMID 40528942
- [Derived] Brunckhorst O, Liszka J, James C, Fanshawe JB, Hammadeh M, Thomas R, Khan S, Sheriff M, Ahmed HU, Van Hemelrijck M, Muir G, Stewart R, Dasgupta P, Ahmed K. Mental wellbeing and quality of life in prostate cancer (MIND-P): Protocol for a multi-institutional prospective cohort study. PLoS One. 2023 Apr 24;18(4):e0284727. doi: 10.1371/journal.pone.0284727. eCollection 2023. PMID 37093833